CLINICAL TRIAL: NCT00696098
Title: Effects of Butyrate on Colonic Health of Patients With Diarrhoea Predominant
Brief Title: Effects of Butyrate on Colonic Health of Patients With Diarrhoea Predominant IBS and UC in Remission
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Top Institute Food and Nutrition (Other)
Responsible Party: Fred Troost, University of Maastricht
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 06-3-067
Record Dates: First submitted 2008-06-09; First posted 2008-06-12 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2009-10

CONDITIONS: Gut Health
MeSH Terms: interventions — Butyric Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): sodium butyrate
  Interventions: Other: sodium butyrate
- 2 (Placebo Comparator)
  Interventions: Other: NaCl

INTERVENTIONS:
Other: sodium butyrate — 1 enema (60 ml) once daily containing 100mM
  Arms: 1
Other: NaCl — 1 enema (60 ml) once daily containing 0.9%NaCl
  Arms: 2

SUMMARY:
Short chain fatty acids (mainly butyrate, acetate, and propionate) are produced in the large intestine by bacterial fermentation of undigested carbohydrates, such as dietary fibres. Butyrate is an important energy source of the intestinal epithelium and has a pivotal role in the regulation of epithelial cell proliferation and differentiation, immune function and mucosal protection.

Non-digestible carbohydrates (prebiotics) increase the concentrations of colonic butyrate, which has been proposed to be responsible for its beneficial effects. Furthermore, butyrate enemas have been proven to be effective in the treatment of active ulcerative colitis.

In the present study, the direct effects of butyrate on inflammation and parameters of colonic defence and mucosal integrity of the distal colon will be studied in 40 patients with diarrhoea predominant IBS (D-IBS) and 40 patients with ulcerative colitis in remission (UCrem) using rectal enemas. These patients groups were chosen because they have a low-grade inflammation in the large intestine, and can therefore be used as a model to study the mechanistic effects of butyrate. The design used to study the effects of butyrate in both patient groups will be a double blind randomized placebo-controlled parallel design.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of UC or Diarrhea predominant IBS
* Stable western diet
* Age between 18 and 65
* BMI between 18 and 35
* Written informed consent

Exclusion Criteria:

* All enemas and suppository during or 2 weeks prior to the study
* Use of corticosteroids during or 1 month prior to the study
* Use of antibiotics during or 3 months prior to the study
* Budesonide during or 2 weeks prior to the study
* Changes in medication during or 1 month prior to the study
* Lactation, pregnancy and planning of pregnancy
* Previous intestinal surgery
* Clinically significant systemic diseases
* Excessive drinking (>20 alcoholic consumptions per week)
* Changes in prebiotic and/or probiotic use during and 2 weeks prior to the study
* Previous radiotherapy or chemotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-05; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
inflammatory parameters | okt 2008

SECONDARY OUTCOMES:
oxidative stress parameters | okt 2008

CONTACTS AND LOCATIONS:
Overall Officials: Fred Troost, PhD, Principal Investigator — Maastricht University
Locations (1):
- University of Maastricht, Maastricht, Limburg, Netherlands